CLINICAL TRIAL: NCT01116414
Title: Molecular Phenotypes for Cystic Fibrosis Lung Disease
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 08-1509; 5R01HL095396 (NIH); 697 (Other: UNC)
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Cystic Fibrosis; Lung Diseases
MeSH Terms: conditions — Cystic Fibrosis; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to develop an integrated view of molecular mechanisms underlying CF lung disease severity.

DETAILED DESCRIPTION:
BACKGROUND:

Cystic fibrosis (CF) is a recessive genetic disorder caused by mutations in CF transmembrane conductance regulator (CFTR) gene. CF has multi-organ involvement, but respiratory disease is the major cause of morbidity and mortality. The median age of survival in CF is only 37 years, but there is a broad range of disease severity in the lung, even among patients with identical CFTR genotypes, including deltaF508 homozygotes.

DESIGN NARRATIVE:

This project holds great promise for defining a robust molecular phenotype for CF lung disease, which relates to prognosis, and new targets for therapy. By using a large and well-defined population of deltaF508 homozygotes who also have whole genome single nucleotide polymorphism (SNP) data, and by studying gene expression across the whole transcriptome in a large number of samples of two relevant tissues (respiratory epithelium and transformed lymphocytes), we will be uniquely positioned to develop an integrated view of molecular mechanisms underlying CF lung disease severity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with CF
* Participation in Genetic Modifiers of CF Lung Disease study (NCT00037765)

Exclusion Criteria:

* History of lung transplant
* Fully anticoagulated or clotting abnormalities
* Large nosebleed in the last 2 months
* Acutely ill

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CF patients who have the same CFTR genetic background, i.e., homozygous deltaF508, and who are at the extremes of pulmonary phenotype, i.e., the most severe and mildest lung disease.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2009-07; Primary Completion 2011-12-13 (Actual); Study Completion 2023-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Knowles, MD, Principal Investigator — University of North Carollina at Chapel Hill
Locations (3):
- United States (3):
  - Johns Hopkins University, Baltimore, Maryland
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Case Western Reserve University, Cleveland, Ohio

REFERENCES:
- [Background] Drumm ML, Konstan MW, Schluchter MD, Handler A, Pace R, Zou F, Zariwala M, Fargo D, Xu A, Dunn JM, Darrah RJ, Dorfman R, Sandford AJ, Corey M, Zielenski J, Durie P, Goddard K, Yankaskas JR, Wright FA, Knowles MR; Gene Modifier Study Group. Genetic modifiers of lung disease in cystic fibrosis. N Engl J Med. 2005 Oct 6;353(14):1443-53. doi: 10.1056/NEJMoa051469. PMID 16207846
- [Background] O'Neal WK, Gallins P, Pace RG, Dang H, Wolf WE, Jones LC, Guo X, Zhou YH, Madar V, Huang J, Liang L, Moffatt MF, Cutting GR, Drumm ML, Rommens JM, Strug LJ, Sun W, Stonebraker JR, Wright FA, Knowles MR. Gene expression in transformed lymphocytes reveals variation in endomembrane and HLA pathways modifying cystic fibrosis pulmonary phenotypes. Am J Hum Genet. 2015 Feb 5;96(2):318-28. doi: 10.1016/j.ajhg.2014.12.022. Epub 2015 Jan 29. PMID 25640674
- [Background] Polineni D, Dang H, Gallins PJ, Jones LC, Pace RG, Stonebraker JR, Commander LA, Krenicky JE, Zhou YH, Corvol H, Cutting GR, Drumm ML, Strug LJ, Boyle MP, Durie PR, Chmiel JF, Zou F, Wright FA, O'Neal WK, Knowles MR. Airway Mucosal Host Defense Is Key to Genomic Regulation of Cystic Fibrosis Lung Disease Severity. Am J Respir Crit Care Med. 2018 Jan 1;197(1):79-93. doi: 10.1164/rccm.201701-0134OC. PMID 28853905
- [Background] Dang H, Polineni D, Pace RG, Stonebraker JR, Corvol H, Cutting GR, Drumm ML, Strug LJ, O'Neal WK, Knowles MR. Mining GWAS and eQTL data for CF lung disease modifiers by gene expression imputation. PLoS One. 2020 Nov 30;15(11):e0239189. doi: 10.1371/journal.pone.0239189. eCollection 2020. PMID 33253230